CLINICAL TRIAL: NCT04167683
Title: The Effect of Medical Treatment on Muscle Dysfunction and the Prognostic Role of Muscle Dysfunction at Critical Decision Points in Patients With Hematological Diseases Referred to Myeloablative Hematopoietic Stem Cell Transplant (HSCT), to Myeloablative HSCT With a "Reduced Toxicity Conditioning" Regime With Fludarabine and Treosulfane (FluTreo), or to Non-myeloablative HSCT. - A Prospective Observational Study.
Brief Title: Muscle Dysfunction in Patients With Hematological Diseases Referred to Stem Cell Transplant
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jan Christensen, post doc, Rigshospitalet, Denmark
Other Study IDs: P-2019-223
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Diseases; Chronic Myeloid Leukemia; Acute Myeloid Leukemia; Acute Lymphoid Leukemia; Myelodysplastic Syndromes; Non Hodgkin Lymphoma; Stem Cell Transplant Complications; Chronic Lymphocytic Leukemia
Keywords: Muscle mass; Muscle strength; Complications; Patient reported outcomes; PRO; Physical function; hematopoietic stem cell transplant
MeSH Terms: conditions — Hematologic Diseases; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Patients referred to myeloablative HSCT: These patients will undergo 5 assessments: a baseline-assessment 3-4 week prior to conditioning treatment, at discharge (in-patients) or at day +28 after stem cell infusion (out-patients) and follow-up assessments at 3 months, 6 months and 12 months.
  Interventions: Other: No intervention
- Cohort 2 - Patients referred to non myeloablative HSCT: These patients will undergo 5 assessments: a baseline-assessment 3-4 week prior to conditioning treatment, at discharge (in-patients) or at day +28 after stem cell infusion (out-patients) and follow-up assessments at 3 months, 6 months and 12 months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
PURPOSE: To investigate the effect of the disease and HSCT on muscle dysfunction and to investigate the prognostic role of muscle dysfunction at critical decision points in patients with hematological diseases referred to hematopoietic stem cell transplant (HSCT).

HSCT: Patients diagnosed with malignant hematological diseases who are referred to myeloablative HSCT, to a myeloablative "reduced toxicity conditioning" regime with Fludarabine and Treosulfane (FluTreo) or to non-myeloablative HSCT.

DETAILED DESCRIPTION:
RATIONAL: Patients diagnosed with malignant hematological diseases undergoing HSCT are faced with poor prognosis. The treatment is demanding and associated with severe deconditioning potentially leading to worse prognostic outcomes. To what extend patients body composition at the point of referral to HSCT, as well as changes in body composition throughout the cancer continuum is associated with cancer outcomes is currently not well described, specifically if this should be part of standard clinical evaluation in order to optimize therapy-efficacy. Recent findings suggest that pathophysiological alterations in skeletal muscle mass and function can have significant implications for the risk of disease progression and long term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute myelogenous leukaemia (AML), acute lymphatic leukaemia (ALL), chronic myelomonocytic leukaemia (CMML), myelodysplastic syndrome (MDS), chronic lymphatic leukaemia (CLL), malignant lymphomas or multiple myeloma (MM) referred to myeloablative HSCT, myeloablative RTC-HSCT or non-myeloablative HSCT at the Department of Haematology, Rigshospitalet, Blegdamsvej.

Exclusion Criteria:

* age <18; pregnancy; physical or mental disabilities precluding test of muscle function; inability to read and understand Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant hematological diseases referred to myeloablative HSCT, myeloablative RTC-HSCT or non-myeloablative HSCT.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 and Cohort 2 Medical treatment complications | From baseline to 1 year follow-up
  Incidens rate of medical complications (mortality, re-hospitalization, infections, all cause disease relapse, chronic GVHD, return to work)

SECONDARY OUTCOMES:
Hospitalization duration | From baseline to 1 year follow-up
  Total number days in hospital
Disease free survival | From baseline to 1 year follow-up
  Risk of disease progression
Overall survival | From baseline to 1 year follow-up
  Risk of mortality from any-cause
Change in whole body lean mass | From baseline to 1 year follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in appendicular lean mass | From baseline to 1 year follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in whole body fat percentage | From baseline to 1 year follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in visceral fat mass | From baseline to 1 year follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in bone mineral density | From baseline to 1 year follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in bone mineral content | From baseline to 1 year follow-up
  Dual-energy X-ray Absorptiometry (DXA) scan
Change in walking capacity | From baseline to 1 year follow-up
  Maximum 10 meter walking speed
Change in lower body physical function | From baseline to 1 year follow-up
  30 seconds Sit-To- Stand test
Change in maximum leg power | From baseline to 1 year follow-up
  Leg extensor power test
Change in inflammation markers | From baseline to 1 year follow-up
  Blood values are registered from the patients hospital record in relation to assessments. C-reactive protein (CRP) and leucocytes are registered as they are inflammation markers
Change in creatinine and hemoglobin | From baseline to 1 year follow-up
  Blood values are registered from the patients hospital record in relation to assessments. C-reactive protein (CRP) and leucocytes are registered as they have an influence on muscle strength
Change in body fat percentage, fat mass, fat-free mass, muscle mass and bone mass and total body water | From baseline to 1 year follow-up
  Bioelectrical Impedance Analyzer
Change in health related quality of life | From baseline to 1 year follow-up
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30 Version 3.0)
Change in psychological distress | From baseline to 1 year follow-up
  Hospital Anxiety and Depression Scale (HADS) questionnaire
Change in sleep quality | From baseline to 1 year follow-up
  Pittsburgh Sleep Quality Index (PSQI) questionnaire
Change in physical activity level | From baseline to 1 year follow-up
  International Physical Activity Questionnaire (IPAQ) short form

CONTACTS AND LOCATIONS:
Overall Officials: Jan Christensen, post doc, Principal Investigator — Department of Occupational- and Physiotherapy, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Not provided